CLINICAL TRIAL: NCT07343583
Title: Effectiveness of Transcutaneous Tibial and Sacral Nerve Stimulation in Preventing the Development of Detrusor Overactivity in Patients With Subacute Suprasacral Spinal Cord Injury
Brief Title: Effects of Sacral and Tibial Stimulation on Bladder Function in Subacute Suprasacral Spinal Cord Injury
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2-25-900
Record Dates: First submitted 2025-12-22; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-12

CONDITIONS: Spinal Cord Injury; Detrusor Overacitivity
Keywords: transcutaneous sacral stimulation; transcutaneous tibial stimulation; detrusor overactivity; neurogenic bowel dysfunction; subacute spinal cord injury
MeSH Terms: conditions — Spinal Cord Injuries; Urinary Bladder, Overactive

STUDY DESIGN:
Intervention Model Description: Participants with subacute suprasacral spinal cord injury will be randomly assigned into three parallel groups.
  One group will receive tibial nerve stimulation, the second group will receive sacral nerve stimulation, and the control group will receive no stimulation.
  Urodynamic outcomes will be compared between the three groups after the intervention period.
  Functional and symptom-based questionnaires will be assessed before the intervention and after urodynamic evaluation, and both within-group and between-group comparisons will be performed.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- transcutaneous tibial nerve stimulation (Active Comparator): Subacute suprasacral spinal cord injury patients receiving transcutaneous tibial nerve stimulation.
  Interventions: Device: Transcutaneous Tibial Nerve Stimulation
- transcutaneous sacral nerve stimulation (Active Comparator): Subacute suprasacral spinal cord injury patients receiving transcutaneous sacral nerve stimulation.
  Interventions: Device: Transcutaneous Sacral Nerve Stimulation
- Control group (No Intervention): Data from patients who have not undergone any stimulation prior to urodynamics in the standard protocol will be used. Urodynamic results will be evaluated by comparing them between groups.

INTERVENTIONS:
Device: Transcutaneous Tibial Nerve Stimulation — For patients in the TTNS group, two adhesive surface electrodes will be placed: the negative electrode immediately behind the right medial malleolus, and the positive electrode 10 cm above the negative electrode along the tibial nerve. The correct position of the negative electrode will be confirmed by the visualization of the flexion of the big toe or toes, which spreads with increasing current intensity. Stimulation will be applied in continuous mode at a frequency of 20 Hz and a pulse duration of 200 msec. The intensity will then be increased to the highest level tolerated by the patient, which will not cause lower extremity muscle spasm in patients with complete SCI and will not cause discomfort in the stimulation areas in patients with incomplete SCI. TTSS sessions will be administered 5 times per week, for a total of 15 sessions, each lasting 30 minutes.
  Arms: transcutaneous tibial nerve stimulation
Device: Transcutaneous Sacral Nerve Stimulation — For the TSNS group, electrodes will be placed symmetrically 5 cm lateral to both sides at the level determined by manual palpation of the sacrum over the S3 foramen, and the current intensity will be increased until contraction is observed in the patient's external anal sphincter. The current frequency will be 20 Hz, the impulse duration will be 200 microseconds, and the treatment will be administered 15 times at 30-minute intervals 5 times a week.
  Arms: transcutaneous sacral nerve stimulation

SUMMARY:
Suprasacral spinal cord injury (SCI) frequently leads to neurogenic detrusor overactivity (NDO), resulting in elevated bladder storage pressures, urinary incontinence, and an increased risk of upper urinary tract damage. Early regulation of bladder function is a key objective of SCI rehabilitation, particularly during the subacute phase when pathological spinal reflex pathways are still developing.

Pharmacological treatments are considered first-line therapy for NDO; however, adequate control may not be achieved in all patients, and treatment tolerance may be limited. Non-invasive neuromodulation techniques have emerged as alternative or adjunctive approaches for managing lower urinary tract dysfunction, but evidence regarding their effectiveness in SCI-related NDO-especially when applied during the subacute period-remains limited.

This prospective randomized comparative study aims to evaluate and compare the effectiveness of transcutaneous sacral neurostimulation (TSNS) and transcutaneous tibial neurostimulation (TTNS) applied during the subacute phase of suprasacral SCI in preventing the development of neurogenic detrusor overactivity. A secondary objective is to assess the effects of these interventions on the severity of neurogenic bowel dysfunction.

Eligible adult patients with subacute suprasacral SCI will be randomized into three groups: TTNS, TSNS, or a control group receiving standard care without neuromodulation prior to urodynamic assessment. Urodynamic parameters including detrusor pressure, bladder compliance, and maximal cystometric capacity, will be compared between groups. Functional outcomes and symptom severity related to neurogenic bladder and bowel dysfunction will also be evaluated.

By investigating non-invasive neuromodulation strategies applied early after SCI, this study aims to contribute evidence regarding the prevention of NDO development and to support the optimization of neuromodulation use in clinical practice for individuals with suprasacral SCI.

DETAILED DESCRIPTION:
Neurogenic detrusor overactivity (NDO) is a common consequence of suprasacral spinal cord injury (SCI) and represents a major risk factor for urinary incontinence and upper urinary tract deterioration. During the subacute phase following SCI, maladaptive spinal reflex pathways associated with detrusor overactivity are still evolving. Interventions applied during this period may influence the development and severity of long-term bladder dysfunction.

Non-invasive neuromodulation techniques have been shown to modulate afferent neural pathways involved in lower urinary tract control. Transcutaneous tibial neurostimulation (TTNS) has demonstrated efficacy in both neurogenic and non-neurogenic bladder dysfunction, while evidence regarding transcutaneous sacral neurostimulation (TSNS) remains limited. Comparative data evaluating these two transcutaneous approaches in subacute SCI-related NDO are lacking.

This prospective randomized comparative study is designed to evaluate the effects of TTNS and TSNS applied during the subacute phase of suprasacral SCI on the prevention of NDO development. Adult patients with traumatic or non-traumatic suprasacral SCI within six months of injury will be enrolled and randomly assigned to one of three groups: TTNS, TSNS, or a control group receiving standard care without neuromodulation prior to urodynamic evaluation.

Participants in the intervention groups will receive non-invasive transcutaneous neuromodulation administered 15 sessions. Following completion of sessions, all groups will undergo standardized urodynamic assessment in accordance with International Continence Society (ICS) recommendations. Urodynamic parameters including maximal detrusor pressure during filling, bladder compliance, and maximal cystometric capacity, will be evaluated and compared between groups.

In addition to urodynamic outcomes, functional status and symptom severity related to neurogenic bladder and neurogenic bowel dysfunction will be assessed using validated clinical scales. A secondary analysis will examine the impact of TTNS and TSNS on the severity of neurogenic bowel dysfunction during the subacute SCI period.

This study aims to clarify the role of early, non-invasive neuromodulation in modulating bladder and bowel dysfunction following suprasacral SCI. The findings are expected to contribute to evidence-based decision-making regarding early intervention strategies and to support the development of standardized transcutaneous neuromodulation protocols in SCI rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18-65 years of age
2. Injury duration <6 months
3. Traumatic and non-traumatic SCI;
4. Patients with spinal cord injury above T11

Exclusion Criteria:

1. Patients with a cardiac pacemaker
2. Patients with other neurological diseases that may affect neurogenic bladder (Parkinson's disease, polyneuropathy, neurodegenerative disease, cerebrovascular disease, etc.)
3. Patients with structural abnormalities in the genitourinary system (pelvic floor dysfunction, BPH, etc.)
4. Patients with acute urinary tract infection
5. Patients with a history of pelvic fracture associated with SCI
6. Patients using medications that may affect NDO (anticholinergic-sympathomimetic, etc.)
7. Patients who have undergone another neuromodulation technique after injury
8. Patients who have previously undergone pelvic radiation, bladder cancer, or other surgical procedures performed on the bladder that may affect bladder physiology will not be included in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-08-05 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of urodynamic data in patients with subacute suprasacral spinal cord injury | A single urodynamic assessment is performed immediately after completion of the 3-week stimulation protocol (no later than 24 hours after the final session) and once for each patient.
  The primary outcome is the comparison of urodynamic parameters among three groups: tibial nerve stimulation, sacral stimulation, and control group without stimulation in patients with subacute suprasacral spinal cord injury

SECONDARY OUTCOMES:
Neurogenic Bladder Dysfunction Score | This measurement will be performed twice. 1. During the initial evaluation of the patient (before stimulation has begun) 2. One month after the completion of urodynamic testing in patients who have completed stimulation
  It is a score specifically developed to assess symptoms and outcomes associated with neurogenic bladder dysfunction. It is a 24-item questionnaire (0-74 points). The higher the score, the greater the severity of symptoms. Its validity and reliability in Turkish have been demonstrated.
Neurogenic Bowel Dysfunction Score | This measurement will be performed twice. 1. During the initial evaluation of the patient (before stimulation has begun) 2. One month after the completion of urodynamic testing in patients who have completed stimulation
  It was developed to assess neurogenic bowel dysfunction in patients with spinal cord injury. It consists of 10 items related to the impaired quality of life caused by bowel symptoms. Its validity and reliability in Turkish have been demonstrated.
Spinal Cord Independence Measure III (SCIM III) | This measurement will be performed twice. 1. During the initial evaluation of the patient (before stimulation has begun) 2. One month after the completion of urodynamic testing in patients who have completed stimulation
  It is specifically designed to cover all aspects related to individuals with SCI, including self-care ability, respiratory and sphincter management, and daily mobility. SCIM results reflect the independence of individuals with SCI; a higher score indicates that very little assistance or fewer helpers are needed to complete basic daily living and life support activities.

CONTACTS AND LOCATIONS:
Overall Officials: Zuhal Özişler, associate professor, Principal Investigator — Ankara City Hospital Bilkent
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fergany LA, Shaker H, Arafa M, Elbadry MS. Does sacral pulsed electromagnetic field therapy have a better effect than transcutaneous electrical nerve stimulation in patients with neurogenic overactive bladder? Arab J Urol. 2017 Mar 29;15(2):148-152. doi: 10.1016/j.aju.2017.01.007. eCollection 2017 Jun. PMID 29071144
- [Result] Stampas A, Gustafson K, Korupolu R, Smith C, Zhu L, Li S. Bladder Neuromodulation in Acute Spinal Cord Injury via Transcutaneous Tibial Nerve Stimulation: Cystometrogram and Autonomic Nervous System Evidence From a Randomized Control Pilot Trial. Front Neurosci. 2019 Feb 19;13:119. doi: 10.3389/fnins.2019.00119. eCollection 2019. PMID 30837835
- [Result] Redshaw JD, Lenherr SM, Elliott SP, Stoffel JT, Rosenbluth JP, Presson AP, Myers JB; Neurogenic Bladder Research Group (NBRG.org). Protocol for a randomized clinical trial investigating early sacral nerve stimulation as an adjunct to standard neurogenic bladder management following acute spinal cord injury. BMC Urol. 2018 Aug 29;18(1):72. doi: 10.1186/s12894-018-0383-y. PMID 30157824
- [Result] Sonmez R, Yildiz N, Alkan H. Efficacy of percutaneous and transcutaneous tibial nerve stimulation in women with idiopathic overactive bladder: A prospective randomised controlled trial. Ann Phys Rehabil Med. 2022 Jan;65(1):101486. doi: 10.1016/j.rehab.2021.101486. Epub 2021 Nov 11. PMID 33429090
- [Result] Yamanishi T, Kaga K, Fuse M, Shibata C, Uchiyama T. Neuromodulation for the Treatment of Lower Urinary Tract Symptoms. Low Urin Tract Symptoms. 2015 Sep;7(3):121-32. doi: 10.1111/luts.12087. Epub 2015 Feb 17. PMID 26663726